CLINICAL TRIAL: NCT00046553
Title: Glucocorticoid and Mineralocorticoid Receptor Function in Post Traumatic Stress Disorder
Brief Title: Brain Receptor Function in Post-Traumatic Stress Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020317; 02-M-0317
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-10

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Cortisol; CRH; HPA Axis; Hypothalamus; Hippocampus; Post-Traumatic Stress Disorder; PTSD; Healthy Volunteer
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mifepristone

INTERVENTIONS:
Drug: RU-486 (Mifepristone)

SUMMARY:
The purpose of this study is to examine the function of cortisol receptors in post-traumatic stress disorder (PTSD).

Patients with PTSD have neurobiological dysregulation of the hypothalamic-pituitary-adrenal (HPA) axis function. High corticotrophin releasing hormone (CRH) levels and decreased hippocampal volume are major features of the disorder. The mechanisms responsible for these alterations are not known. This study will evaluate the function of cortisol receptors to determine their roles in maintaining PTSD HPA axis dysregulation. Three groups of subjects will take part in the study: Patients with PTSD, healthy control subjects who were exposed to trauma in the past and remained healthy and healthy control subjects who were never traumatized

At study entry, the cerebral spinal fluid (CSF) of all participants will be sampled and evaluated. Participants will also undergo a magnetic resonance imaging (MRI) scan of the brain as well as eye blink trace conditioning and neuropsychological tests.

Participants will be admitted to the Clinical Center for two nights on three different occasions. At each overnight visits, blood levels of stress hormones will be measured every hour for 26 hours after medication or placebo are given. This will be the end of the study for both groups of healthy control subjects, with the exception that they may be asked to repeat neuropsychologic and eye blink tests after 12 weeks.

Participants with PTSD will receive paroxetine for 10 weeks. After 10 weeks these participants will be reevaluated in exactly the same way as before treatment (except they will not repeat the MRI scan).

DETAILED DESCRIPTION:
We propose to investigate the underlying mechanisms that account for neurobiological dysregulation of HPA axis function in PTSD. Paradoxically, low or normal plasma and urinary cortisol despite high corticotrophin releasing hormone (CRH) levels are a major feature of this disorder. Some investigators report decreased hippocampal volume in patients with PTSD. The mechanisms responsible for these alterations are not known. One possibility is that patients with PTSD have an increased number of glucocorticoid receptors (GR) and/or increased GR sensitivity, causing hyper-suppression of HPA axis. Another possibility is that high CRH levels lead to increased mineralocorticoid receptor (MR) levels and this up-regulation of MR is responsible for the low cortisol secretion seen in PTSD. Elevated CRH levels could also result in reduced hippocampal volume.

In order to evaluate MR and GR function, we will examine the effect of RU486 (Mifepristone; a GR antagonist), spironolactone (Aldactone; an MR antagonist), and placebo, on cortisol and ACTH plasma levels in patients with PTSD, trauma exposed, and non-trauma exposed healthy controls. The extent of increase in cortisol and/or ACTH after administration of antagonists will reflect the inhibition ordinarily imposed by GR and MR. We will also examine subjects' cerebral spinal fluid (CSF), CRH levels, and hippocampal volume. Following this evaluation, patients with PTSD will be treated with paroxetine for 8 weeks. The assessments performed before treatment will then be repeated.

The first aim of the present study is to elucidate the pathophysiology of PTSD through the examination of the roles of GR and MR in maintaining PTSD HPA axis dysregulation. The second aim is to compare CSF CRH levels across groups in an effort to extend previous findings and determine whether CRH levels in PTSD are higher than levels in trauma exposed healthy subjects. The present investigation will also evaluate the relationship between CRH levels in PTSD, MR/GR function, hippocampal volume and hippocampally-mediated cognitive tasks. Finally, we will examine the effects of long-term paroxetine treatment in PTSD on HPA axis function, hippocampal volume, and hippocampally-mediated cognitive tasks.

ELIGIBILITY:
INCLUSION CRITERIA:

18 to 65 years of age.

Male and female.

Score greater than or equal to 50 on the Clinician-Administered PTSD Scale (CAPS-2) as a baseline measure of PTSD symptom severity.

Capable of providing informed consent, obtained prior to any study procedures.

Free of all psychotropic medication for at least 2 weeks, excluding short-term hypnotics. Patients who were treated with fluoxetine will only be included after a medication free period of at least 8 weeks.

Good physical health, confirmed by a complete physical exam (including normal vital signs), electrocardiogram, neurologic exam, and routine laboratory tests of blood and urine. However, if patients have participated in other research studies or have had blood work through their primary MD within the last 6 months, these results will be used instead of repeating blood draws for inclusion into the study.

EXCLUSION CRITERIA:

Patients who meet DSM-IV criteria for substance abuse (alcohol or drugs) or substance dependence within 6 months prior to screening. The effect of abuse/dependence on phenomenology and biology could mask and exceed PTSD effect.

Patients at current risk for homicide or suicide.

All additional DSM IV Axis I comorbidity, excluding secondary diagnoses of major depressive disorder (MDD) or anxiety disorder (AD). Given the high comorbidity of these disorders in PTSD, and since excluding such patients would not provide the full spectrum of the disorder, only patients in whom axis I diagnoses of MDD and AD preceded onset of PTSD will be excluded.

Pregnant women (all stages) and women of childbearing potential who are not practicing a clinically accepted method of contraception or who have a positive pregnancy test or who are lactating.

Blood donation (1 Red Cross Unit) within the 8 weeks preceding the study. This is the minimal safe period between consecutive donations.

Subjects who are doing well on medication. Although we will only recruit non-medicated patients, the decision to stop medication will be taken purely on clinical grounds. No subject will be taken off medication solely to participate in the study.

Unable to comply with study procedures or assessments as regards the screening evaluation (i.e. PTSD diagnosis, health requirements, etc.) and the 3 hospitalization for evaluation of glucocorticoid and mineralocorticoid receptor function.

Subjects who are allergic to mifepristone, paroxetine or spironolactone, and subjects with any contraindication to treatment with these agents (as described in their current labeling), will be excluded from participation in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 97
Dates: Start 2002-09; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Yehuda R. Biology of posttraumatic stress disorder. J Clin Psychiatry. 2001;62 Suppl 17:41-6. PMID 11495096
- [Background] Gesing A, Bilang-Bleuel A, Droste SK, Linthorst AC, Holsboer F, Reul JM. Psychological stress increases hippocampal mineralocorticoid receptor levels: involvement of corticotropin-releasing hormone. J Neurosci. 2001 Jul 1;21(13):4822-9. doi: 10.1523/JNEUROSCI.21-13-04822.2001. PMID 11425909
- [Background] Bremner JD, Randall P, Scott TM, Bronen RA, Seibyl JP, Southwick SM, Delaney RC, McCarthy G, Charney DS, Innis RB. MRI-based measurement of hippocampal volume in patients with combat-related posttraumatic stress disorder. Am J Psychiatry. 1995 Jul;152(7):973-81. doi: 10.1176/ajp.152.7.973. PMID 7793467